CLINICAL TRIAL: NCT00113984
Title: Phase I Trial of a PSA Based Vaccine and an Anti-CTLA-4 Antibody in Adults With Metastatic Androgen Independent Prostrate Cancer
Brief Title: Vaccine and Antibody Treatment of Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050167; 05-C-0167; NCT00124670 (obsolete NCT alias)
Record Dates: First submitted 2005-06-11; First posted 2005-06-13 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2012-11-07

CONDITIONS: Prostatic Neoplasms
Keywords: Monoclonal Antibody; Vaccine; Cytokines; Immunotherapy; Elispot Assay; Prostate Cancer; Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ipilimumab; sargramostim

INTERVENTIONS:
Biological: PROSTVAC-V/TRICOM
Biological: PROSTVAC-F/TRICOM
Drug: MDX-010
Drug: Sargramostim

SUMMARY:
This study will evaluate the side effects of a fixed dose of vaccine and GM-CSF with increasing doses of anti-CTLA-4 antibody in patients with advanced prostate cancer. The vaccine consists of a "priming vaccine" called PROSTVAC/TRICOM, made from vaccinia virus, and a "boosting vaccine" called PROSTVAC-F/TRICOM, made from fowlpox virus. GM-CSF is a chemical that boosts the immune system, and anti-CTLA-4 antibody is a protein that may improve anti-tumor activity and the response to the vaccines. DNA is inserted into the priming and boosting vaccine viruses to cause production of proteins that enhance immune activity and also to produce prostate specific antigen (PSA)-a protein that is normally produced by the patient's tumor cells.

Patients 18 years of age and older with androgen-insensitive prostate cancer that has spread beyond the original site may be eligible for this 7-month study. Candidates must have disease that has worsened despite treatments with hormones and up to one chemotherapy regimen. Their tumor must produce PSA, and they must have no history of allergy to eggs or egg products Candidates are screened with a medical history and physical examination, blood and urine tests, electrocardiogram, pathological confirmation of the diagnosis and presence of the PSA marker, chest x-rays, imaging studies to assess the extent of tumor, and, if clinically indicated, a cardiologic evaluation.

Participants receive the priming vaccination on study day 1. After 2 weeks and then again every 4 weeks while on the study, they receive a boosting vaccine. All vaccines are injected under the skin. On the day of each vaccination and daily for the next 3 days, patients receive an injection of GM-CSF to increase the number of immune cells at the vaccination site. On the day of the first six boosting vaccinations, they receive anti-CTLA-4 antibody as an infusion through a vein over 90 minutes.

Patients are monitored for safety and treatment response with the following tests and procedures:

* Blood and urine tests monthly, or more often if needed, to monitor liver, kidney, and other organ function.
* Imaging studies to assess the tumor before starting treatment, again around study days 99 and 183, and then every 3 months after that while on study.
* Apheresis (a procedure for collecting immune cells called lymphocytes) to measure the immune response to treatment. Apheresis is done three times: before starting the study and again around study days 99 and 183. For this procedure, blood is collected through a needle in an arm vein. The blood circulates through a machine that separates it into its components by spinning, and the lymphocytes are extracted. The rest of the blood is returned to the patient through the same needle. This will only be done in participants who have the tissue marker HLA-A2 (about 50% of patients).

Patients whose disease responds to treatment and who do not develop severe side effects may continue treatment beyond the initial 7-month study period on vaccine alone (without the antibody). After treatment is completed, patients are monitored for up to 15 years. This includes a medical history and physical examination for 5 years following the last vaccination. Information beyond 5 years is collected once a year by telephone.

DETAILED DESCRIPTION:
Background:

* Adenocarcinoma of the prostate is the most common cancer diagnosis in American males, and the second leading cause of cancer death.
* The proposed vaccine strategy represents a third-generation design that elicits a T-cell immune response to cells expressing PSA and has been shown to break tolerance to this self-antigen, and cause objective response and PSA declines in patients with metastatic AIPC.
* This strategy also utilizes an antibody to CTLA-4 that may block the normal signals to down regulate the immune response following active vaccination.
* Anti CTLA-4 antibodies have been associated with autoimmune events that are generally manageable and have been associated with clinical response.

Objectives:

* To determine the safety and tolerability of a combination of a fixed dose of vaccine and anti-CTLA4, which will be dose escalated.
* To evaluate immunologic response (as measured by an increase in PSA specific T-cells measured by ELISPOT in HLA-A2+ patients), and clinical response (as measured by RECIST and PSA consensus criteria).

Eligibility:

* Must have metastatic androgen insensitive prostate cancer with no bone pain requiring narcotics and have had no more prior chemotherapy.
* Life expectancy greater than or equal to 6 months. ECOG 0-1
* Should have no autoimmune diseases; no evidence of being immunocompromised; no serious intercurrent medical illness; no cardiac disease; no prior splenectomy.
* No prior treatment with MDX-010 (Ipilimumab).
* No brain metastasis, history of seizures, encephalitis, or multiple sclerosis.
* No serious hypersensitivity reaction to egg products.

Design:

* This is an open label, phase I safety trial with sequential cohorts of patients all receiving a fixed dose of PSA-TRICOM vaccines and sargramostim, with dose escalation of MDX-010 (Ipilimumab).
* PROSTVAC -V/TRICOM (vaccinia) 2 x 10(8) pfu subcutaneously will be administered as the initial priming vaccine on day 1 of cycle 1 only.
* PROSTVAC -F/TRICOM (fowlpox) 1 x 10(9) pfu subcutaneously starting on day 15 followed by monthly boosting vaccination. Sargramostim 100 mcg per day will be administered subcutaneously at the vaccination site on days 1-4 of each vaccine cycle (prime and boost).
* MDX-010 (Ipilimumab) will be administered, as per the assigned dose level, as a 90-minute intravenous infusion on the same day as the monthly boosting vaccinations with PROSTVAC-F/TRICOM (fowlpox). After 6 courses of MDX-010, patients may receive Maintenance dose of MDX-010 every 3 months until there is evidence of disease progression or toxicity, for up to an additional 12 months (equivalent to 4 additional MDX-010 courses).
* Monthly boosting vaccinations with PROSTVAC-F/TRICOM (fowlpox) and sargramostim may then continue until patients meet off study criteria.

ELIGIBILITY:
* INCLUSION CRITERIA:

A. Histopathological documentation of prostate cancer confirmed in the Laboratory of Pathology at the: NIH Clinical Center, National Institutes of Health (NIH), the National Naval Medical Center, or Walter Reed Army Medical Center prior to starting this study. If no pathologic specimen is available, patients may enroll with a pathologist's report showing a histologic diagnosis of prostate cancer and a clinical course consistent with the disease.

B. Must have metastatic androgen insensitive prostate cancer with no bone pain requiring narcotics and have had no prior chemotherapy.

C. Life expectancy greater than or equal to 6 months.

D. ECOG performance status of 0-1.

E. No systemic steroid or steroid eye drop use within 2 weeks prior to initiation of experimental therapy.

F. Hematological eligibility parameters

* Granulocyte count greater than or equal to1,500/mm(3)
* Platelet count greater than or equal to100,000/mm(3)
* Hgb greater than or equal to 9 Gm/dL
* Lymphocyte count greater than or equal to 500/mm(3).

G. Biochemical eligibility parameters (within 16 days of starting therapy)

-Hepatic function: Bilirubin less than or equal to 1.5 mg/dl (OR in patients with Gilbert's syndrome, a total bilirubin less than or equal to 3.0 mg/dL), AST and ALT less than or equal to 2.5 times upper limit of normal

H. No other active malignancies within the past 12 months (with the exception of non-melanoma skin cancers or carcinoma in situ of the bladder) or life threatening illnesses.

I. Willing to travel to the NIH for follow-up visits.

J. 18 years of age or greater.

K. Vaccinia-naive or vaccinia immune.

L. Able to understand and sign informed consent.

M. Agree to use adequate contraception prior to study entry and for at least 4 months following the last vaccine injection.

N. Patients must remain on medical castration therapy, unless they have had surgical castration

O. Patients must have recovered from acute toxicities related to prior therapy or surgery. For chemotherapy typically this is 3-4 weeks.

P. Parameters for assessment of baseline renal function:

* Serum creatinine not above the institution limits of normal, OR creatinine clearance on a 24 hour urine collection of greater than or equal to 60 mL/min.
* Patients must have less than grade 2 proteinuria (unless the cause is determined not to be renal.)

EXCLUSION CRITERIA:

A. Patients should have no evidence of being immunocompromised as listed below.

* Human immunodeficiency virus positivity due to the potential for decreased tolerance and may be at risk for severe side effects.
* Hepatitis B or C positivity
* Concurrent use of topical steroids (including steroid eye drops) or systemic steroids. Nasal or inhaled steroid use is permitted

B.Patients should have no autoimmune diseases that have required treatment such as, Addison's disease, Hashimoto's thyroiditis, or systemic lupus erythematous, Sjogren syndrome, scleroderma, Goodpasture syndrome, and active Grave's disease. Also excluded are patients with autoimmune hemolytic anemia, ulcerative and hemorrhagic colitis, endocrine disorders (e.g., thyroiditis, hyperthyroidism, hypothyroidism, autoimmune hypophysitis/hypopituitarism, and adrenal insufficiency), sarcoid granuloma, myasthenia gravis, polymyositis, and Guillain-Barre syndrome. Patients with a history of autoimmunity that has not required systemic immunosuppressive therapy or does not threaten vital organ function including CNS, heart, lungs, kidneys, skin, and GI tract will be allowed.

C. History of allergy or untoward reaction to prior vaccination with vaccinia virus or to any component of the vaccinia vaccine regimen.

D. Do not administer the recombinant vaccinia vaccine if the recipient, or for at least three weeks after vaccination, their close household contacts (close household contacts are those who share housing or have close physical contact) are: persons with active or a history of eczema or other eczematoid skin disorders; those with other acute, chronic or exfoliative skin conditions (e.g., atopic dermatitis, burns, impetigo, varicella zoster, severe acne, or other open rashes or wounds) until condition resolves; pregnant or nursing women; children 3 years of age and under; and immunodeficient or immunosuppressed persons (by disease or therapy), including HIV infection.

E. Serious intercurrent medical illness (e.g., one that requires treatment) which would interfere with the ability of the patient to carry out the treatment program, including, but not limited to, inflammatory bowel disease, Crohn's disease, ulcerative colitis, or active diverticulitis.

F. Patients with cardiac disease that have fatigue, palpitation, dyspnea or angina with ordinary physical activity (New York Heart Association class 2 or greater) are not eligible.

G. Patients with a history of congestive heart failure or who have objective evidence of congestive heart failure by physical exam or imaging are not eligible.

H. Patients with pulmonary disease that have fatigue or dyspnea with ordinary physical activity are not eligible.

I. Concurrent chemotherapy.

J. No brain metastasis, or with a history of seizures, encephalitis, or multiple sclerosis.

K. Serious hypersensitivity reaction to egg products.

L. Prior splenectomy.

M. Patients who have received prior MDX-01.

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-06-08; Primary Completion 2008-02-01 (Actual); Study Completion 2011-12-01 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of a combination of a fixed dose of vaccine and anti-CTLA4, which will be dose escalated.

SECONDARY OUTCOMES:
To evaluate immunologic response (as measured by an increase in PSA specific T-cells measured by ELISPOT in HLA-A2+ patients), and clinical response (as measured by RECIST and PSA consensus criteria).

CONTACTS AND LOCATIONS:
Overall Officials: James L Gulley, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Madan RA, Mohebtash M, Arlen PM, Vergati M, Rauckhorst M, Steinberg SM, Tsang KY, Poole DJ, Parnes HL, Wright JJ, Dahut WL, Schlom J, Gulley JL. Ipilimumab and a poxviral vaccine targeting prostate-specific antigen in metastatic castration-resistant prostate cancer: a phase 1 dose-escalation trial. Lancet Oncol. 2012 May;13(5):501-8. doi: 10.1016/S1470-2045(12)70006-2. Epub 2012 Feb 10. PMID 22326924
- [Background] Gulley JL, Dahut WL. Future directions in tumor immunotherapy: CTLA4 blockade. Nat Clin Pract Oncol. 2007 Mar;4(3):136-7. doi: 10.1038/ncponc0749. No abstract available. PMID 17327854
- [Background] Theoret MR, Arlen PM, Pazdur M, Dahut WL, Schlom J, Gulley JL. Phase I trial of an enhanced prostate-specific antigen-based vaccine and anti-CTLA-4 antibody in patients with metastatic androgen-independent prostate cancer. Clin Genitourin Cancer. 2007 Jun;5(5):347-50. doi: 10.3816/CGC.2007.n.017. No abstract available. PMID 17645835